CLINICAL TRIAL: NCT01931046
Title: A Phase 1 / 2a Study of In-situ REIC/Dkk-3 Therapy in Patients With Localized Prostate Cancer (MTG-REIC-PC003)
Brief Title: Use of Recombinant Adenovirus Therapy to Treat Localized Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Momotaro-Gene Inc. (Industry)
Collaborators: The Pacific Link Consulting Co (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MTG-REIC-PC003
Record Dates: First submitted 2013-08-21; First posted 2013-08-29 (Estimated); Last update posted 2020-09-04 (Actual); Status verified 2020-09

CONDITIONS: Localized Prostate Cancer
Keywords: prostate cancer; adenocarcinoma of the prostate
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Masking Description: open label
Oversight: Data Monitoring Committee: No

ARMS (2):
- Part 1 (Experimental): Treatment at one of three dose levels of Ad5-SGE-REIC/Dkk-3 in a sequential dose-escalating design with 4 cycles of therapy at each dose level permitted.
  Interventions: Drug: Ad5-SGE-REIC/Dkk3
- Part 2 (Experimental): Treatment with Ad5-SGE-REIC/Dkk-3 every 6-weeks for up to 4 cycles of therapy and may continue therapy if they have stable disease or are responding.
  Interventions: Drug: Ad5-SGE-REIC/Dkk3

INTERVENTIONS:
Drug: Ad5-SGE-REIC/Dkk3 — Ad5-SGE-REIC/Dkk-3, was designed to increase intracellular production REIC protein. The adenovirus vector is a transport mechanism to infuse the REIC protein into the cell providing a temporary transfusion of protein that induces apoptosis in target cancer cells, but does not appear to have a significant effect on normal tissues.

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of AD5-SGE-REIC/Dkk-3 in patients with localized prostate cancer.

DETAILED DESCRIPTION:
This is a phase 1/2a clinical trial in subjects who are diagnosed with prostate cancer to evaluate the effectiveness of Ad5-SGE-REIC/Dkk-3 in the treatment of localized prostate cancer.

Subjects enrolled will be diagnosed with localized prostate cancer (clinical stage T1/T2) having a Gleason score of 6 to 7 (3+4 or 4+3). Subjects will receive up to four (4) transrectal ultrasound (TRUS)-guided IT treatments with Ad5-SGE-REIC/Dkk-3 into the prostate approximately 6-weeks apart. Each treatment cycle will be performed using a minimum of three track injections through the prostrate using a total of 3 mL volume. Approximately 2 mL of the total volume will be injected into the most dense areas of cancer based on biopsy and MRI mapping (fusion biopsy) and 1 mL total volume will be injected into the opposite lobe of the prostate or other areas to ensure complete saturation of the prostate over multiple injections.

Subjects who, in the opinion of the investigator, are progressing at any time after the second injection of Ad5-SGE-REIC/Dkk-3 may be discontinued and will be treated according to standard medical practice.

ELIGIBILITY:
Inclusion Criteria:

Key Inclusion Criteria:

Subjects must meet all of the following criteria to be included:

1. Male aged between 50 and 80 years (inclusive) with histologically documented clinically localized, adenocarcinoma of the prostate.
2. Subject with clinical stage T1 or T2 with Gleason score of 6 or 7 (3+4 or 4+3).
3. At least one (1) MRI evaluable tumor with volume of 400 mm3 or greater.
4. At least total of 10 mm of cancer tissue based on an MRI guided 12-core biopsy.
5. Recent (≤ 6 months prior to study entry) negative bone scan and computerized tomography (CT) scan of abdomen/pelvis.
6. Life expectancy of at least 5 years.
7. Subjects should have adequate bone marrow function defined as an absolute peripheral granulocyte count ≥ 1,500 and platelet count of ≥ 100,000, adequate hepatic function with a bilirubin ≤ 1.5 mg/dl and serum glutamic-pyruvic transaminase (SGPT) < 4x the upper limits of normal, adequate renal function defined as serum creatinine ≤ 2.0 mg/dl
8. Subjects must have a coagulation profile (prothrombin time [PT], partial thromboplastin time [PTT]) not more than 2-times the upper limit of normal and no history of substantial non-iatrogenic bleeding diatheses. Use of anticoagulants within 5-days of the Ad5-SGE-REIC/Dkk-3 injections is limited to local use only (for control of central line patency).
9. Subject is willing to refrain from sexual activity or agrees to use a barrier contraceptive device (e.g. condom) for 8-weeks after treatment with Ad5-SGE-REIC/Dkk-3.
10. Subjects must sign an informed consent indicating that they are aware of the investigational nature of the study.

Key Exclusion Criteria

Subjects meeting any of the following criteria will be excluded:

1. Prior primary radiation treatment to the prostate.
2. Severe bladder outlet obstructive disorder (AUA >25) or urinary track retention.
3. Chemotherapy, immunotherapy or other investigational study drug within the past 4 weeks.
4. Unable to tolerate TRUS.
5. Subjects with uncontrolled cardiac, hepatic, renal or neurologic/psychiatric disorders, that in the opinion of the investigator put the subject at significant risk, are not eligible.
6. Subjects who are HIV positive or have active hepatitis B or C infections are not eligible.
7. Subjects with a clinical history of primary or secondary immunodeficiency, autoimmune disease or subjects taking immunosuppressive drugs such as corticosteroids continuously for > 4 months [> 5 mg hydrocortisone/day] are ineligible.
8. As a result of medical review, physical examination, the Principal Investigator (or medically qualified nominee) considers the subject unfit for the study.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2013-10; Primary Completion 2018-07-06 (Actual); Study Completion 2020-03 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose | Up to 24 weeks
  To define the Maximum Tolerated Dose (MTD) or Maximum Feasible Dose (MFD) for intratumoral injection (IT) of Ad5-SGE-REIC/Dkk-3 viral vector.

SECONDARY OUTCOMES:
Effectiveness of Ad5-SGE-REIC/Dkk-3 | Up to 78 weeks
  To assess the effectiveness of Ad5-SGE-REIC/Dkk-3 in the treatment of prostate cancer as evaluated by biomarkers, transrectal ultrasound (TRUS), biopsy and MRI.
Rate and intensity of adverse reactions after treatment with Ad5-SGE-REIC/Dkk-3 | Up to 54 weeks
  To assess the rate of adverse events and grade of adverse events after in-situ therapy with Ad5-SGE-REIC/Dkk-3 protein in prostate cancer subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher J Kane, MD, Principal Investigator — University of California, San Diego; Brian J Miles, MD, FACS, Principal Investigator — Baylor College of Medicine and Methodist Hospital
Locations (3):
- United States (3):
  - UCSD Moores Cancer Center, San Diego, California
  - Brigham and Women's Hospital, Boston, Massachusetts
  - The Methodist Hospital Research Institute, Houston, Texas